CLINICAL TRIAL: NCT07033650
Title: Evaluation of Clinical Performance of Bulk Fill Resin Composite Restorations Using Snow Plow Versus Oscillating Packing Technique: Randomized Controlled Clinical Trial
Brief Title: Evaluation of Clinical Performance of Bulk Fill Resin Composite Restorations Using Snow Plow Versus Oscillating Packing Technique
Acronym: RCT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Suez Canal University (Other)
Responsible Party: Principal Investigator, Basma hosny, Lecturer of Conservative Dentistry, Faculty of Dentistry, Suez Canal University, Suez Canal University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 906/2024
Record Dates: First submitted 2025-04-22; First posted 2025-06-24 (Actual); Last update posted 2025-06-24 (Actual); Status verified 2025-04

CONDITIONS: Caries Class Ii

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control (Active Comparator): teeth will be restored with the packable Bulk-fill composite (X-tra Fil) with a single increment of 4 mm starting with the proximal boxes and cured for 10 s
  Interventions: Other: Bulk-fill composite (X-tra Fil)
- Snowplow" technique (Experimental): teeth will be restored using Snowplow technique where a 1 mm layer of flowable Bulk-fill composite (X-tra Base) will be deposited at the gingival margin of the prepared teeth and kept uncured. Then pushing a heavily filled packable nanohybrid resin composite (X-tra Fil) into the uncured flowable composite.
  The combined layer of flowable and restorative composites will be then cured using LED curing unit for 10 s
  Interventions: Other: Bulk-fill composite (X-tra Fil); Other: flowable Bulk-fill composite (X-tra Base)
- Oscillating technique (Experimental): teeth will be restored using oscillating technique where the packable Bulk-fill composite material will be placed in bulk to fill the prepared cavity using a plastic filling instrument then the compothixo oscillating packing instrument will be used The oscillation energy (140 Hz) will be applied for 30 s, during which the composite will be adapted to all the cavity walls, and then light cured for 10 s.
  Interventions: Other: Bulk-fill composite (X-tra Fil); Device: compothixo oscillating packing

INTERVENTIONS:
Other: Bulk-fill composite (X-tra Fil) — Bulk fill resin composite
Other: flowable Bulk-fill composite (X-tra Base) — flowable resin composite
  Arms: Snowplow" technique
Device: compothixo oscillating packing — oscillating packing device
  Arms: Oscillating technique

SUMMARY:
This is a randomized, controlled, double-blinded clinical trial (the patient and the examiners are blind to the group assignment). Eligible patients will be examined clinically and radiographically using bite-wing radiography, and recruited according to the previously mentioned inclusion and exclusion criteria. All participants will sign written informed consents after being completely aware of the aim, settings, procedures, benefits and potential side effects of the study. Each tooth will be assigned by a number; R1 (Bulk fill RC), R2 (Snow plow tech) and R3 (Oscillating tech). Restoration numbers will be concealed in an opaque sealed envelope that will be held by a facilitator who will not involve in any of the phases of the clinical trial. Every patient will choose an envelope for each tooth. Patients and examiners will be blinded to the material assignment; the operator also will be blinded for the type of restoration during tooth preparation and will be informed only at the time of restoration placement.

Each case will be evaluated according to FDI criteria, based on both functional (Fracture of material and retention, Marginal adaptation, Occlusal contour and wear, Proximal contact point and food impaction, and Radiographic examination) and biological (Postoperative sensitivity, Recurrence of caries and Tooth integrity) properties. Bitewing radiographs and intra-oral photographs will be also used for assessment of all restorations.

Assessment of postoperative sensitivity and tooth vitality will be carried out on the patient by application of a cold stimulus (e.g. a blast of cold air). Postoperative sensitivity will be recorded at the time of restoration placement, and throughout all follow-up appointments, and include type of pain, discomfort and duration, and/or on stimulus at clinical assessment and should always be compared with the response of adjacent vital teeth. Intensity will be assessed also with a visual analogue scale (VAS) which is a commonly used tool for measuring pain.

On a scale of 1 to 5, restorations will be rated as follows; score 1: clinically excellent/very good, 2: clinically good, 3: clinically satisfactory, 4: clinically unsatisfactory but repairable and 5: clinically poor/irrepairable and in need of replacement. So the scores 1, 2 and 3 considered clinically successful while scores 4 and 5 considered clinically not successful.

DETAILED DESCRIPTION:
This is a randomized, controlled, double-blinded clinical trial (the patient and the examiners are blind to the group assignment). The approval of Ethical committee of the Faculty of Dentistry, Suez Canal University, will be taken. This study will be carried on apparently healthy patients of age group 21-50 years, with at least three occluso-proximal cavitated dentinal lesion on the posterior molars, the patients who will agree to participate in this study will sign an informed consent. Also it will be reported according to the protocol established by CONSORT guidelines to ensure transparent and complete reporting.

Patients will be recruited from outpatient clinic of Operative Dentistry Department in Faculty of Dentistry, Suez Canal University. Eligible patients will be examined clinically and radiographically using bite-wing radiography, and recruited according to the previously mentioned inclusion and exclusion criteria. All participants will sign written informed consents after being completely aware of the aim, settings, procedures, benefits and potential side effects of the study. The data from the study and consent forms will be written in Arabic so that every patient could understand them. Patients will be only admitted to the study after signing the informed consent.

Simple randomization will be assigned for 29 participants. Every patient will be diagnosed by examiners for three posterior class II carious lesions. Each tooth will be assigned by a number; R1 (Bulk fill RC), R2 (Snow plow tech) and R3 (Oscillating tech). Restoration numbers will be concealed in an opaque sealed envelope that will be held by a facilitator who will not involve in any of the phases of the clinical trial. Every patient will choose an envelope for each tooth. Patients and examiners will be blinded to the material assignment; the operator also will be blinded for the type of restoration during tooth preparation and will be informed only at the time of restoration placement.

Each case will be evaluated according to FDI criteria, based on both functional (Fracture of material and retention, Marginal adaptation, Occlusal contour and wear, Proximal contact point and food impaction, and Radiographic examination) and biological (Postoperative sensitivity, Recurrence of caries and Tooth integrity) properties. Assessment of restorations will be performed clinically by visual inspection using magnification loupes (4.5x; Carl Zeiss GmbH, Jena, Germany), dental mirrors, a light source and FDI recommended probes with different tip diameters of 150 and 250 micrometer diameter (150x and 250x, Deppeler, Switzerland) . These probes will be used specially for evaluation of both marginal adaptation (functional property) and tooth integrity of enamel cracks and tooth fractures (biological property). Bitewing radiographs and intra-oral photographs will be also used for assessment of all restorations.

Assessment of postoperative sensitivity and tooth vitality will be carried out on the patient by application of a cold stimulus (e.g. a blast of cold air). Postoperative sensitivity will be recorded at the time of restoration placement, and throughout all follow-up appointments, and include type of pain, discomfort and duration, and/or on stimulus at clinical assessment and should always be compared with the response of adjacent vital teeth. Transient pain brought on by stimulation will be acceptable, while persistent pain renders the restoration unacceptable and necessitates intervention to resolve the problem. Intensity will be assessed also with a visual analogue scale (VAS) which is a commonly used tool for measuring pain.

On a scale of 1 to 5, restorations will be rated as follows; score 1: clinically excellent/very good, 2: clinically good, 3: clinically satisfactory, 4: clinically unsatisfactory but repairable and 5: clinically poor/irrepairable and in need of replacement. So the scores 1, 2 and 3 considered clinically successful while scores 4 and 5 considered clinically not successful.

ELIGIBILITY:
Inclusion Criteria:

* Each patient should have at least three occluso-proximal carious lesions in the posterior molars in three different quadrants (two upper and one lower)
* Only co-operative patients approving to participate in the trial.

Exclusion Criteria:

* Patients with disabilities or severe medically compromised.
* Patients with severe bruxism, clenching or temporomandibular joint disorders.
* Patients with allergy to any components of the materials.

Ages: 21 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 87 (Actual)
Dates: Start 2024-01-25 (Actual); Primary Completion 2025-02-02 (Actual); Study Completion 2025-03-21 (Actual)

PRIMARY OUTCOMES:
Adaptation of restorations | at baseline (immediately after restoration), after 3 months, 6 months, and 12 months
  magnifying loupes (4.5x; Carl Zeiss GmbH, Jena, Germany) will be recommended for evaluation. In addition, a set of blunt explorers, straight and double angled for proximal sites, with different blunt tips of 50, 150, and 250 μm will be utilized to assess the gap size between tooth and restoration. The explorer was drawn across the restoration's surface toward the tooth to detect marginal ditching, irregularities or fracture. If the explorer catches, it means the restoration's edges haven't adapted closely to the tooth structure
Radiographic examination of the restorations | at baseline (immediately after restoration), after 3 months, 6 months, and 12 months
  A scale of 5 pints 1-5 , where 1 consider no pathology with harmonious transition between tooth and restoration 2 mean small visible but acceptable excess or gap 3 means gaps or excess still within acceptable range 4 means gaps or marked excess material in inter radicular 5 means gaps or secondary caries or apical pathology or fracture
postoperative sensitivity and tooth vitality using VAS | at baseline (immediately after restoration), after 3 months, 6 months, and 12 months
  Intensity will be assessed also with a visual analogue scale (VAS) which is a tool widely used to measure pain. The Visual Analogue Scale (VAS) consists of a 100 mm horizontal line with the endpoints defining extreme limits such as 'no pain at all' and 'pain as bad as it could be'. The patient is asked to mark his pain level on the line between the two endpoints. Using a ruler, the score was determined by measuring the distance (mm) on the 10-cm line between the "no pain" anchor and the patient's mark, providing a range of scores from 0-100. Score less than 5 mm will be labeled as no pain, scores from 5 to 44 mm will be labeled as mild pain, scores from 45 to 74 mm will be labeled as moderate pain, and scores 75 mm and greater will be labeled as sever pain.

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Dentistry, Suez Canal University, Ismailia, Egypt

IPD SHARING:
Plan to Share IPD: No